CLINICAL TRIAL: NCT04467983
Title: Abaloparatide Added to Ongoing Denosumab vs Continued Denosumab Alone
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Radius Health, Inc. (Industry); Crozer-Keystone Health System (Other)
Responsible Party: Principal Investigator, Joseph Lane, MD, Principal Investigator, Hospital for Special Surgery, New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-1296
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: denosumab; abaloparatide
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Denosumab; abaloparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Denosumab alone (Active Comparator): 3 injections of Denosumab at appropriate times, separated by no more than 7 months from the last treatment.
  Interventions: Drug: Denosumab Injection
- Combination therapy (Active Comparator): 3 injections of Denosumab at appropriate times, separated by no more than 7 months from the last treatment, with added abaloparatide 80 mcg subcutaneously daily, started within 6 months of the last denosumab treatment, for a total of 18 months.
  Interventions: Drug: Denosumab Injection; Drug: Abaloparatide

INTERVENTIONS:
Drug: Denosumab Injection — Denosumab alone: 3 injections of Denosumab at appropriate times, separated by no more than 7 months from the last treatment.
  Other Names: Prolia
Drug: Abaloparatide — Combination therapy: 3 injections of Denosumab at appropriate times, separated by no more than 7 months from the last treatment, with added abaloparatide 80 mcg subcutaneously daily, started within 6 months of the last denosumab treatment, for a total of 18 months.
  Other Names: Tymlos
  Arms: Combination therapy

SUMMARY:
This randomized open label clinical trial will evaluate the effect of continued denosumab alone over 18 months versus denosumab with added abaloparatide for 18 months. 70 postmenopausal women will be enrolled over a period of 18 months. The co-primary outcomes will be group differences in bone mineral density (BMD) of the total hip and lumbar spine at 18 months. Secondary outcomes will include group differences in bone mineral density (BMD) at the femoral neck, trochanter and wrist sites at 6, 12 and 18 months, spine and total hip bone mineral density (BMD) at 6 and 12 months and trabecular bone score (TBS) at 18 months. Secondary outcomes will also include within group changes from baseline for each of these variables. Bone turnover markers will also be measured to demonstrate that PINP levels will increase with administration of abaloparatide even in the setting of ongoing denosumab, while CTX levels will remain low.

DETAILED DESCRIPTION:
Some women on denosumab treatment for osteoporosis remain at high risk for fracture. These include women who sustain incident fractures on denosumab and those who have declining bone mineral density (BMD) or persistently low bone mineral density (BMD), despite treatment. There are few options available for these patients. Denosumab withdrawal is associated with dramatic increased bone remodeling, rapid prominent bone loss, and multiple vertebral fractures (Cummings JBMR 2017). Switching from denosumab to teriparatide is associated with substantial BMD loss in the hip and femoral neck. After 2 years of denosumab treatment, when women are switched to teriparatide, total hip BMD remains below the baseline (at end of denosumab treatment) over the entire 2 years of teriparatide treatment (Leder Lancet 2015).

Abaloparatide might be a better option than teriparatide in patients switching from denosumab, because it is less pro-resorptive than teriparatide, however, hip BMD will still likely decline. Alternatively, adding abaloparatide to ongoing denosumab might be an excellent treatment option for these women. One of the investigators has previously shown that adding teriparatide to ongoing alendronate results in improved BMD and bone strength, compared to switching to teriparatide (Cosman JCEM 2009 and Cosman JBMR 2013). Others have shown that co-administration of teriparatide and denosumab to treatment naïve women increases BMD more than either agent alone (Tsai Lancet 2013, Leder et al JCEM 2014). Based on both of these observations, the investigators believe that adding abaloparatide to continued denosumab treatment will allow bone formation to increase, without increasing bone resorption (modeling-based bone formation) and will produce substantial BMD increments in both spine and hip.

Hypothesis: In women who still appear to be at high risk for fracture while receiving ongoing denosumab therapy, adding abaloparatide will increase BMD of the lumbar spine and total hip significantly more than continuing denosumab alone.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal woman >age 45 of any racial origin
* Participants will have received at least 4 prior denosumab treatments and be within 7 months from their last denosumab injection
* Participants are willing to participate for the duration of the study and have no physical or psychological illness that would prohibit them from participating.
* Diagnosis of osteoporosis based on bone mineral density and/or fracture criteria. Osteoporosis will be defined by bone mineral density T-Score < -2.5 at lumbar spine (at least 2 evaluable vertebrae between L1 and L4), total hip or femoral neck. Osteoporosis will also be defined clinically in women with osteoporotic fractures within the preceding 5 years, including clinical vertebral or nonvertebral fractures or vertebral fracture confirmed by radiograph or lateral DXA VFA image, along with a DXA BMD T-Score < -1.5 at one or more skeletal sites.

Exclusion Criteria:

* Use of drugs other than denosumab (within the preceding 3 months) known to affect skeletal or calcium homeostasis.
* Fewer than 2 evaluable lumbar vertebrae
* A history of a symptomatic renal stone within the past 2 years or history of multiple symptomatic renal stones within the preceding 10 years
* Skeletal Disorders other than osteoporosis, including hypercalcemia, hyperparathyroidism, or Paget's Disease
* History of external or internal radiation therapy
* Estimated GFR below 30 ml/min
* Any contraindications to receipt of Abaloparatide or Denosumab
* History of any cancer in past 5 years (except basal/squamous skin cancer)
* Unexplained elevation of Serum Alkaline Phosphatase
* History of atypical femoral fracture

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density changes at total hip and lumbar spine | 18 months
  Group differences in BMD increment at total hip and lumbar spine at 18 months.

SECONDARY OUTCOMES:
Bone mineral density changes in increments | 6, 12, 18 months
  Group Differences in BMD increments:
  of lumbar spine and total hip at 6 and 12 months. of femoral neck, and 1/3 radius at 6, 12 and 18 months.
  Group Differences in BMD increments:
  of lumbar spine and total hip at 6 and 12 months. of femoral neck, and 1/3 radius at 6, 12 and 18 months.
  Group Differences in BMD increments:
  of lumbar spine and total hip at 6 and 12 months. of femoral neck, and 1/3 radius at 6, 12 and 18 months. Group differences in BMD increments of lumbar spine and total hip (at 6 and 12 months) and of femoral neck and 1/3 distal radius (at 6, 12, and 18 months)
Trabecular Bone Score changes | 18 months
  Group differences in Trabecular Bone Score at 18 months
Within Group Increments in bone mineral density (vs baseline) | 6, 12, 18 months
  Within Group Increments in bone mineral density vs baseline of lumbar spine (at 6, 12, and 18 months) and of total hip, femoral neck, and distal 1/3 radius (at 6, 12, and 18 months)
Differences in biochemical bone turnover markers | 3, 6, 12, 18 months
  Within and between group differences in biochemical bone turnover markers (P1NP and CTX) at 3, 6, 12, and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeri W Nieves, PhD, Study Director — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leder BZ, Tsai JN, Uihlein AV, Wallace PM, Lee H, Neer RM, Burnett-Bowie SA. Denosumab and teriparatide transitions in postmenopausal osteoporosis (the DATA-Switch study): extension of a randomised controlled trial. Lancet. 2015 Sep 19;386(9999):1147-55. doi: 10.1016/S0140-6736(15)61120-5. Epub 2015 Jul 2. PMID 26144908
- [Background] Cosman F, Wermers RA, Recknor C, Mauck KF, Xie L, Glass EV, Krege JH. Effects of teriparatide in postmenopausal women with osteoporosis on prior alendronate or raloxifene: differences between stopping and continuing the antiresorptive agent. J Clin Endocrinol Metab. 2009 Oct;94(10):3772-80. doi: 10.1210/jc.2008-2719. Epub 2009 Jul 7. PMID 19584192
- [Background] Cosman F, Keaveny TM, Kopperdahl D, Wermers RA, Wan X, Krohn KD, Krege JH. Hip and spine strength effects of adding versus switching to teriparatide in postmenopausal women with osteoporosis treated with prior alendronate or raloxifene. J Bone Miner Res. 2013 Jun;28(6):1328-36. doi: 10.1002/jbmr.1853. PMID 23281041
- [Background] Leder BZ, O'Dea LS, Zanchetta JR, Kumar P, Banks K, McKay K, Lyttle CR, Hattersley G. Effects of abaloparatide, a human parathyroid hormone-related peptide analog, on bone mineral density in postmenopausal women with osteoporosis. J Clin Endocrinol Metab. 2015 Feb;100(2):697-706. doi: 10.1210/jc.2014-3718. Epub 2014 Nov 13. PMID 25393645
- [Background] Leder BZ, Tsai JN, Uihlein AV, Burnett-Bowie SA, Zhu Y, Foley K, Lee H, Neer RM. Two years of Denosumab and teriparatide administration in postmenopausal women with osteoporosis (The DATA Extension Study): a randomized controlled trial. J Clin Endocrinol Metab. 2014 May;99(5):1694-700. doi: 10.1210/jc.2013-4440. Epub 2014 Feb 11. PMID 24517156